CLINICAL TRIAL: NCT04939376
Title: Association Between Uterine , Intracavitary , Cervical and Cervical Canal Lesions With in Vitro Fertilization/Intracytoplasmic Sperm Injection(IVF/ICSI) Outcome.
Brief Title: Uterine Lesions and Their Association to Invitro Fertilization(IVF) or Intracytoplasmic Sperm Injection(ICSI) Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mostafa Ahmed, doctor, Assiut University
Other Study IDs: Uterine lesions and ICSI
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Women with hysteroscopically or ultrasonographic detected uterine anomalies(adenomyosis,fibroid) intracavitary lesions ( like polyp, adhesion or septum) and those with detected endometrial abnormalities (like hypervascularization,pale endometrium) ,cervical lesion and cervical canal lesion or pelvic lesion
  Interventions: Procedure: IVF
- Group B: Matched women (eg. Age,parity, BMI, ovarian reserve….) with no uterine or ovarian abnormalities assessed by hysteroscopy or ultrasonography.
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: IVF — In vitro fertilization

SUMMARY:
1. To study the effect of uterine wall , intracavitary , cervical as well as cervical canal lesion on the outcome of IVF/ICSI cycle.
2. To establish a score for prediction of IVF/ICSI cycle success .

DETAILED DESCRIPTION:
IVF is one of the most successful treatment of fertility, (1) however, several IVF cycles fail to achieve pregnancy (2).failure defined as three or more failed attempts of ICSI (3). Implantation failure is a complex in nature, may be due to structural or functional causes (3, 4).

that previously undiagnosed, misinterpreted initial diagnoses, or subtle newly added intrauterine abnormalities may be a significant cause of IVF failure (5, 6), studies say that intra-uterine pathologies represent 40-50 % of causes of ICSI failure (7, 8), hysteroscopic removal of endometrial polyps, submucous fibroids, uterine septum, or intrauterine adhesions could increase the pregnancy rate (9). so, Evaluation of the uterine cavity may become a routine investigation before assisted reproductive technology(ART) procedures (10).

In this study, we evaluate the relationship between the different uterine and cervical pathologies and decreased live birth rate.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 38 years old.

  * An indication for IVF/ICSI..
  * Women with BMI between 18.5 : 29.9 .
  * Women with normal antimullerian hormone(AMH), antral follicle count(AFC) (good responders).

Exclusion Criteria:

Refusal to join the study.

* Women with age less than 18 and more than 38 .
* Women with BMI less than 18.5 and more than 30 .
* Untreated tubal hydrosalpinges.
* Poor responders as assessed by AFC 4 or less ,AMH O.8 ng/dl (nice 2013).

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women between 18 and 38 years old.
  * An indication for IVF/ICSI..
  * Women with BMI between 18.5 : 29.9 .
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | Baseline
  Pregnancy rate with IVF/ICSI with uterine lesions

CONTACTS AND LOCATIONS:
Overall Officials: Momen Kamel, Prof.dr, Study Director — Assiut University

REFERENCES:
- [Background] Rai R, Regan L. Recurrent miscarriage. Lancet. 2006 Aug 12;368(9535):601-11. doi: 10.1016/S0140-6736(06)69204-0. PMID 16905025
- [Background] Dicker D, Ashkenazi J, Feldberg D, Farhi J, Shalev J, Ben-Rafael Z. The value of repeat hysteroscopic evaluation in patients with failed in vitro fertilization transfer cycles. Fertil Steril. 1992 Oct;58(4):833-5. doi: 10.1016/s0015-0282(16)55338-2. PMID 1426335
- [Background] Levi Setti PE, Colombo GV, Savasi V, Bulletti C, Albani E, Ferrazzi E. Implantation failure in assisted reproduction technology and a critical approach to treatment. Ann N Y Acad Sci. 2004 Dec;1034:184-99. doi: 10.1196/annals.1335.021. PMID 15731311